CLINICAL TRIAL: NCT07395336
Title: Elacestrant and Exemestane for Patients With Pretreated HR+/HER2- Metastatic Breast Cancer and [18F] FES-avid Lesions (COMBINE): a Proof-of-concept Phase 2 Clinical Trial
Brief Title: Elacestrant and Exemestane for Patients With Pretreated HR+/HER2- Metastatic Breast Cancer and [18F] FES-avid Lesions (COMBINE)
Acronym: COMBINE-01
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UID 4270
Record Dates: First submitted 2025-12-05; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
Keywords: elacestrant; exemestane; HR+; HER2-
MeSH Terms: conditions — Breast Neoplasms | interventions — elacestrant; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- elacestrant and exemestane (Experimental): elacestrant 345 mg die and exemestane 25 mg die
  Interventions: Drug: elacestrant and exemestane

INTERVENTIONS:
Drug: elacestrant and exemestane — elacestrant 345 mg die and exemestane 25 mg die

SUMMARY:
Single agent endocrine therapy (ET), with selective estrogen receptor degraders (SERDs; i.e. fulvestrant or elacestrant), is an option for patients with pre-treated hormone receptor-positive (HR+) breast cancer (BC) with indolent behaviour beyond the first line therapy with CDK4/6 inhibitors (CDK4/6i) + ET, in order to spare the adverse events related to chemotherapy.

Anyway, the efficacy of endocrine monotherapy in patients progressing on first line therapy is low, because of the occurrence of endocrine resistance mechanisms, like the HR loss and the switch to HR-negative subtype, caused by the selective pressure of first line therapy; furthermore, biomarkers for patient selection are missing.

Recently, the 16a-[18F]fluoro-17b-estradiol positron emission tomography ([18F]FES-PET) demonstrated a sensitivity and specificity of 86% in estrogen receptor expression prediction; therefore it is a promising tool to select patients progressing on CDK4/6i + ET without HR loss.

Single agent endocrine therapy (ET), with selective estrogen receptor degraders (SERDs; i.e. fulvestrant or elacestrant), is an option for patients with pre-treated hormone receptor-positive (HR+) breast cancer (BC) with indolent behaviour beyond the first line therapy with target cyclin-dependent kinases 4 and 6 inhibitors (CDK4/6i) + ET, in order to spare the adverse events related to chemotherapy.

Anyway, the efficacy of endocrine monotherapy in patients progressing on first line therapy is low, because of the occurrence of endocrine resistance mechanisms, like the Hormon Receptor (HR) loss and the switch to HR-negative subtype, caused by the selective pressure of first line therapy; furthermore, biomarkers for patient selection are missing.

Recently, the 16a-[18F] fluoro-17b-estradiol positron emission tomography ([18F] FES-PET) demonstrated a sensitivity and specificity of 86% in estrogen receptor expression prediction; therefore it is a promising tool to select patients progressing on CDK4/6i + ET without HR loss.

The combination of endocrine agent, namely fulvestrant 250 mg plus anastrozole 1 mg (an aromatase inhibitor), demonstrated to provide an overall survival benefit in patients with Hormon Receptor positive Breast Cancer only in first line setting but not in patients progressing to ET. However, meanwhile, fulvestrant 500 mg was demonstrated to be superior to fulvestrant 250 mg in 2nd line setting, and oral SERDs (e.g. Elacestrant, Camizestrant) were demonstrated to be superior in terms of Progression Free Survival to fulvestrant 500 mg in patients progressing on ET, in the subgroup of patients with estrogen receptor 1 gene (ESR1) mutations.

Hypothesis: there is a strong rationale to assess the safety and the activity of Elacestrant plus exemestane in patients with pre-treated HR+ and Human Epidermal Growth Factor Receptor 2 negative (HER2-) metastatic breast cancer and at least 50% of [18F]FES-avid measurable lesions, using [18F]FES PET/CT to evaluate the early response to treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Must be at least 18 years old;
2. Must have a histologically- or cytologically-proven diagnosis of carcinoma of the breast with evidence of either locally advanced disease not amenable to resection or radiation therapy with curative intent or metastatic disease not amenable to curative therapy
3. Must be appropriate candidates for endocrine therapy (no visceral crisis, highly symptomatic disease or rapidly progressing disease)
4. Must have 1 of the following as defined by RECIST v1.1:

   1. Measurable disease
   2. Bone only disease with evaluable lesions. Subjects must have at least 1 lytic or mixed lytic/blastic bone lesion; blastic lesions only are not evaluable and allowed. Subjects who have had prior radiation to bone must have at least 1 evaluable lesion in a nonirradiated area.
5. ≥50% of measurable lesions defined as avid (SUVmax≥1.5) at 18F-FES-PET/CT;
6. Must have HR+ and HER2- disease at the last previous biopsy. ER and HER2 testing must be performed in the following manner:

   1. Documentation of ER+ tumor with ≥ 10% staining by immunohistochemistry (IHC), with or without PgR positivity AND
   2. Documentation of HER2- tumor with an IHC result of 0 or 1+ for cellular membrane protein expression or an in situ hybridization negative result as defined in the 2023 ASCO recommendations for HER2 testing (Wolff, 2013; Wolff, 2018; Wolff 2023)

8. Must have progressed during or within 28 days of completion of prior treatment with a CDK4/6 inhibitor in combination with anastrozole or letrozole (+ LHRH agonist for male or premenopausal female patients).

1. This treatment has to be received in first line setting for metastatic disease (with abemaciclib, ribociclib or palbociclib)
2. Discontinuation of prior CDK4/6 inhibitor due to toxicity, in the absence of progression, will not fulfill this criterion
3. Patients must have received the combination treatment for at least 12 months and there must have been evidence of disease control (stable disease [SD], partial response [PR] or complete response [CR] as best response) 9. Must have received no other treatment after the CDK4/6 inhibitor combined with endocrine therapy 10. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1

Exclusion Criteria:

1. Prior treatment with fulvestrant, elacestrant or investigational SERD or ER antagonist in metastatic or early disease (e.g., D-0502, GDC-0810, GDC-0927, GDC-9545, G1T-48, LSZ102, AZD9496, SAR439859, ZN-c5, H3B-6545, bazedoxifene, lasofoxifene)
2. Prior treatment with tamoxifen or SERD alone or combined with CDK4/6i in metastatic setting
3. Any other endocrine therapy < 14 days before first dose of study drug
4. Any prior treatment after first line with CDK4/6i in metastatic setting
5. Bisphosphonates or RANKL inhibitors initiated or dose changed < 3 months prior to first dose of study drug
6. Radiation therapy within 14 days (28 days for brain lesions) before the first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
6-month Progression Free Survival (PFS) rate per RECIST (Response Evaluation Criteria in Solid Tumors) v1.1 | 6 month

SECONDARY OUTCOMES:
Adverse Event (AE) per Common Terminology Criteria for Adverse Events (CTCAE) 5.0 | up to 3 years
Median Overall Survival (OS) | up to 3 years
Overall Response Rate (ORR) per RECIST v1.1 | up to 3 years
Median QoL (QLQ-C30) change from baseline to week 8 of treatment | up to 8 weeks
  Median QoL change from baseline to week 8 of treatment measured by EORTC QLQ-C30 av.4 questionarie
Median QoL (FACT-ES) change from baseline to week 8 of treatment | up to 8 weeks
  Median QoL change from baseline to week 8 of treatment measured by EORTC FACT-ES v.4 questionarie
6-months Progression Free Survival (PFS) rate per RECIST v1.1 according to baseline FES-SUV and SUV variation of FES | 6 months

OTHER OUTCOMES:
6-months Progression Free Survival (PFS) rate per RECIST 1.1 by ESR1/PIK3CA mutation, ER≥50%/PgR≥50% expression, APOBEC+/HRD+/PAM-50 luminal status | 6 month
Progression Free Survival (PFS) rate per RECIST v1.1 by genomic and epigenomic alterations at baseline and after 4 weeks of treatment | up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Curigliano, Principal Investigator — European Institute of Oncology

IPD SHARING:
Plan to Share IPD: No